CLINICAL TRIAL: NCT06607510
Title: Exercise in Patients With Atrial Fibrillation: Effect of Different Types of Exercise on the Burden of the Pathology, on the Biochemical Profile, and on the Functional Capacity of the Patients.
Brief Title: Exercise Effects on Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-DOC004-AF
Record Dates: First submitted 2024-02-22; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation
Keywords: HIFT; HIIT; Intervallic training; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Prospective single-center randomized clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The evaluators of the patients and the person analysing the data will be blinded to the patient's group allocation and te corresponding codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental HIIT. (Experimental): Subjects belonging to this group perform a 12-week supervised exercise. Treadmill walking exercise. Participants must complete four four-minute blocks at an intensity of 85-95% of peak heart rate.
  Interventions: Other: Experimental HIIT
- Experimental HIFT. (Experimental): Subjects belonging to this group perform a 12-week supervised exercise. Four blocks of 4 minutes each of the highest number of repetitions/rounds possible (AMRAP) at an intensity of 85-95% of peak heart rate.
  Interventions: Other: Experimental HIFT
- No intervention: Control. (No Intervention): These patients do not receive training sessions.

INTERVENTIONS:
Other: Experimental HIIT — Subjects belonging to this group perform a 12-week supervised exercise (3 sessions weekly spaced at least 48 hours apart with a maximum duration of 40 minutes), followed by 12 weeks of detraining follow-up. Before starting the intervention, two familiarization sessions for assessing strength and functional capacity will be conducted. This program is designed in a standardized warm-up: joint mobility exercises and neuromuscular activation (5 minutes). Main part os the training is design in treadmill walking exercise (28 minutes). Participants must complete four four-minute blocks at an intensity of 85-95% of peak heart rate.The initial starting speed is 5 km/h and adjust the intensity with incline increments of 2%. Between sets, a prescribed active rest period lasts three minutes, during which patients walk on the treadmill at an intensity of 60-70% of peak heart. The last part of the training is a cool-down (5 minutes treadmill walking at an intensity of 50-60% of peak heart rate).
  Arms: Experimental HIIT.
Other: Experimental HIFT — Subject belonging to this group perform a 12-week supervised exercise (3 sessions weekly spaced at least 48 hours apart with a maximum duration of 40 minutes), followed by 12 weeks of detraining follow-up. Before starting the intervention, two familiarization sessions for assessing strength and functional capacity will be conducted. AMRAP will consist of a circuit of six global, functional exercises with external loads [i) squat; ii) rowing; iii) dead weight; iv) chest press; v) step up; vi) farmer walk]. Patients will perform 10 repetitions of each exercise and complete as many rounds as possible within the specified time. Between blocks, there will be a prescribed active rest period lasting three minutes, during which patients will walk on the treadmill at an intensity of 60-70% of peak heart rate. The last part of the training is a cool-down (5 minutes treadmill walking at an intensity of 50-60% of peak heart rate).
  Arms: Experimental HIFT.

SUMMARY:
Atrial fibrillation (AF) significantly affects quality of life and increases the demand for medical care of those affected. It is very important to identify triggering factors, such as oxidative stress or N-terminal pro-B-type natriuretic peptide (NT-proBNP), as well as to identify potential biomarkers through plasma analysis. At the same time, it is essential to establish adequate training and rehabilitation programs, which would result in a decrease in hospitalizations and the health care costs associated with the pathology. Current cardiac rehabilitation programs based on physical exercise, especially moderate intensity continuous training (MICT), have demonstrated effectiveness. MICT improves cardiorespiratory fitness and quality of life in patients with AF. However, high-intensity intervallic training (HIIT) has shown superior benefits in these variables.

Although HIIT traditionally has an aerobic focus, a variant called high-intensity functional training (HIFT) is suggested that incorporates muscle strengthening exercises recommended in the guidelines for AF management. This innovative modality seeks to achieve cardiovascular and neuromuscular adaptations simultaneously, with a high transfer to daily activities. Despite its potential, the effects at the functional, molecular and clinical levels in patients with AF are unknown. The purpose of the study is to determine the benefits of HIFT on molecular, functional and clinical variables in patients with AF, and to compare these benefits with those achieved with HIIT and the usual care and recommendations in current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation.
* Age between 18 and 80 years.
* Sedentary lifestyle.
* Signed informed consent.

Exclusion Criteria:

* Permanent atrial fibrillation.
* Moderate to severe left ventricular dysfunction.
* Moderate to severe left valvulopathy.
* Severe pulmonary hypertension.
* Ischemic heart disease with incomplete revascularization.
* Arrhythmogenic cardiomyopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of proteins in blood (proteome). | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Venous blood samples are collected from the antecubital vein and kept at 4°C until preparation to avoid clotting and minimise protein degradation. Samples are centrifuged at 1500 g for 10 minutes at 4°C.
  Samples shall are stored at -80°C for subsequent analysis and only one freeze-thaw cycle shall be allowed. All samples shall are prepared within 1 hour of sample collection and show no signs of haemolysis.
  The protein concentrarion will be analyzed (μg/ml).
Oxidative stress status | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Oxidative stress is measured through the analysis of plasma oxidative stress biomarkers concentrations in pg/ml.
Cardiac function: concentrations (pg/ml) of NT-proBNP (type B natriuretic peptide). | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Measurement of cardiac dysfunction is analyzed through the presence of plasma markers of cardiac injury (NT-proBNP; pg/ml).
Maximal strength of upper and lower extremity muscles. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Maximal strength of upper and lower extremity muscles from one concentric repetition maximum (1RM) of half squat and bench press will be assessed (maximal strength).
  Measurements in weight lifted and the number of times. Maximum Repetition or 1RM is the maximum weight (kg) you can move in just one time.
Functional variables: power strength by bar displacement | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in bar displacement in centimeter (cm).
Functional variables: power strength by propulsive velocity | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Mean propulsive velocity (in meter per second).
Functional variables: power strength | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Average power (in watts).
Functional variables: Handgrip strength. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in the manual dynamometer measurements (in kg).
Functional variables: Assessment of cardiorespiratory capacity. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in measurements by a treadmill. The following variables will be assessed before and after the cardiorespiratory capacity measurement:
  1. Gas exchange analysis (VO2, VCO2), in ml·kg-1·min-1.
  2. Maximum speed in treadmill (km/h).
  3. Blood pressure (systolic pressure and diastolic pressure in mm Hg).
  4. Heart rate (bpm).
  5. Rate of perceived exertion (RPE) using a RPE-CR10 scale.
Functional variables: Assessment of functional capacity (6MWT). | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in six-minute walk test (6MWT): number of laps around the hallway and the additional distance covered on the last lap if it is not completed using the markings in the hallway. The outcome measure is quantified in meters.
Functional variables: Levels of physical activity | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  GT3X+ accelerometers estimate physical activity levels based on the accelerometer output in units called "counts per minute".
Clinical variables: Short Form-36 Health Survey (SF-36). | 0 weeks, 13 weeks, 24 weeks.
  The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). A final item, termed self-reported health transition, is answered by the client but is not included in the scoring process. The SF-36 offers a choice of recall format at a standard (4 week) or acute (1 week) time frame. Likert scales and yes/no options are used to assess function and well-being on this 36-item questionnaire. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value.
Clinical variables: Atrial fibrillation burden. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in electrocardiogram (electrical signal from the heart to detect different heart conditions).
Clinical variables: Atrial fibrillation burden (subjective measurement). | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in Atrial Fibrillation Effect on Quality-of-life (AFEQT) questionnaire: palpitations, dyspnea, fatigue and limitations in daily activities. AFEQT evaluates health-related quality of life (HRQoL) and provides an overall score; plus scores for symptoms, daily activities, treatment concerns, and treatment satisfaction.
  20 questions on 7-point Likert scale Overall or subscale scores range from 0-100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).
Clinical variables: Arterial stiffness. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in the images of the right common carotid artery are obtained using an ultrasound.
Clinical variables: Heart rate variability. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  Changes in the variation in the time intervals between heartbeats (R-R intervals).
Clinical variables: Vascular dysfunction. | 0 weeks, 2 weeks, 13 weeks, 24 weeks.
  The cardio-ankle vascular index (CAVI) is a new index of the overall stiffness of the artery from the origin of the aorta to the ankle. CAVI values range from 3 to 18. Depending on the cut-off values.
  Standardized values established by the manufacturer, a value < 8 is considered normal, between 8 and 9 is borderline, and 9 is high and indicates advanced atherosclerosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea Miguel de Cervantes, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No